CLINICAL TRIAL: NCT00174187
Title: Treatment With Recombinant Human Growth Hormone Genotonorm (Registered) in Children With Short Stature Secondary to a Long Term Corticoid Therapy. A Study of Efficacy and Safety.
Brief Title: Treatment With Recombinant Human Growth Hormone (GH) in Children With Short Stature Secondary to a Long Term Corticoid Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-MET-9002-0009; A6281016
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Endocrine System Diseases
MeSH Terms: conditions — Endocrine System Diseases | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatropin (Experimental)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — liquid, daily, until final height Dosage: 0,46 mg/kg/week . The maximum dose should not exceed 50 µg/Kg/day

SUMMARY:
* To assess the effect of a long-term treatment by Genotonorm on linear growth in children with short stature receiving steroid therapy
* To assess the effect of a long term treatment with Genotonorm on bone mineralisation
* To assess the effect of a long term treatment with Genotonorm on body composition

DETAILED DESCRIPTION:
This trial terminated on 10-Jun-2011 due to prolonged issues with drug accountability and data collection discrepancies. The decision to terminate was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Children with juvenile arthritis or nephrotic syndrome
* Before or during puberty

Exclusion Criteria:

* Diabetes Type 1 and 2
* Endocrine disease, except well substituted hypothyroidism

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2000-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Paris, France

REFERENCES:
- [Derived] David H, Aupiais C, Louveau B, Quartier P, Jacqz-Aigrain E, Carel JC, Simon D. Growth Outcomes After GH Therapy of Patients Given Long-Term Corticosteroids for Juvenile Idiopathic Arthritis. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4578-4587. doi: 10.1210/jc.2017-01455. PMID 29029101
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=307-MET-9002-0009&StudyName=Treatment%20with%20Recombinant%20Human%20Growth%20Hormone%20%28GH%29%20in%20Children%20with%20Short%20Stature%20Secondary%20to%20a%20Long%20Term%20Corticoid%20Therap

RESULTS

PARTICIPANT FLOW:
Groups:
- Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis): Participants with juvenile idiopathic arthritis (JIA) received somatropin (Genotropin, Genotonorm) 1.4 International Units per kilogram per week (IU/kg/week), equivalent to 0.46 milligram/kg/week (mg/kg/week), divided in 7 daily doses subcutaneously for up to 3 years. After treatment for 3 years, participants in this group were assigned to Somatropin- After Year 3 group.
- Somatropin- Up To Year 3 (Nephrotic Syndrome): Participants with nephrotic syndrome (NeS) received somatropin (Genotropin, Genotonorm) 1.4 IU/kg/week, equivalent to 0.46 mg/kg/week, divided in 7 daily doses subcutaneously for up to 3 years. After treatment for 3 years, participants in this group were assigned to Somatropin- After Year 3 group.
- Somatropin- After Year 3: Participants with JIA/NeS, who consented to receive treatment beyond 3 years, received somatropin (Genotropin, Genotonorm) 1.4 IU/kg/week, equivalent to 0.46 mg/kg/week divided in 7 daily doses subcutaneously until the additional study drug dose evaluation visit and thereafter received somatropin (Genotropin, Genotonorm) up to 50 microgram (mcg)/kg/day subcutaneously until the final height (FH) was reached or up to Year 11. Final height was confirmed to have been achieved if the growth velocity was less than or equal to 1.5 centimeter (cm) per year during the preceding 12 months and bone age was greater than or equal to 17 years for boys and 15 years for girls.
Period: Period 1 (up to 3 Years)
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome) | Somatropin- After Year 3
Started | 15 | 15 | 0
Completed | 15 | 11 | 0
Not Completed | 0 | 4 | 0
Not completed — Serious adverse event | 0 | 1 | 0
Not completed — Non compliance | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0
Period: Between Period 1 and Period 2
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome) | Somatropin- After Year 3
Started | 0 | 0 | 26
Consented | 0 | 0 | 24
Completed | 0 | 0 | 21
Not Completed | 0 | 0 | 5
Not completed — Did not consent to continue treatment | 0 | 0 | 2
Not completed — Consented, not assigned to treatment | 0 | 0 | 3
Period: Period 2 (After 3 Years)
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome) | Somatropin- After Year 3
Started | 0 | 0 | 21
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 11.14 (3.32) | 11.96 (3.80) | 11.55 (3.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 6 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Height Standard Deviation Score According to Chronological Age (SDS/CA) at Year 3
Description: Height was measured using a wall mounted device (example, Harpenden stadiometer). Height SDS/CA was obtained by measuring the height, subtracting chronological age- and gender-appropriate mean height and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 3
Population: Full Analysis Set (FAS) up to Year 3: included all participants who had at least 1 post-baseline height measurement and were treated with the study drug for at least 1 year.
Measure: Median (Inter-Quartile Range); unit: Standard Deviation Score (SDS)
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
Standard Deviation Score (SDS)
  Baseline | -3.6 [-5.1 to -2.3] | -2.5 [-2.8 to -2.2]
  Change at Year 3 | 0.2 [-1.5 to 1.8] | 1.1 [0.8 to 1.5]

2. Primary Outcome: Change From Baseline in Height Standard Deviation Score According to Chronological Age (SDS/CA) at Final Height
Description: as for outcome 1
Time Frame: Baseline, when final height was reached (assessed up to Year 11)
Population: FAS- after Year 3: included all participants who received at least 1 dose of the study treatment and who had at least 1 post-baseline height measurement. Here, 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin- After Year 3
Number analyzed (Participants) | 21
SDS
  Baseline (n = 21) | -2.86 [-5.61 to -1.00]
  Change at Final Height (n = 4) | 0.71 [0.27 to 3.08]

3. Primary Outcome: Change From Baseline in Weight Standard Deviation Score (SDS) at Final Height
Description: Body weight was measured using a balance scale. Weight SDS was obtained by measuring the weight, subtracting age- and gender-appropriate mean weight and dividing the result by standard deviation of that mean (as obtained from age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, when final height was reached (assessed up to Year 11)
Population: FAS- after Year 3: included all participants who received at least one dose of the study treatment and who had at least one post-baseline height measurement. Here, 'n' signifies those participants who were evaluable for this measure at given time point.
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin- After Year 3
Number analyzed (Participants) | 21
SDS
  Baseline (n = 21) | -1.53 [-4.77 to 2.64]
  Change at Final Height (n = 4) | -0.43 [-1.37 to 1.09]

4. Primary Outcome: Puberty Stage at Final Height
Description: Pubertal stage (graded from I to V for breast development and pubic hair development) according to the Tanner's method was collected. A low stage (Stage I) corresponds to a pre-pubertal stage and a high stage (Stage V) to an adult stage.
Time Frame: When final height was reached (assessed up to Year 11)
Population: FAS- after Year 3: included all participants who received at least one dose of study treatment and who had at least one post-baseline height measurement. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n'=participants who were evaluable for given components of puberty assessment.
Measure: Number; unit: participants
Arm/Group | Somatropin- After Year 3
Number analyzed (Participants) | 4
participants
  Pubic hair: Stage I (n=4) | 0
  Pubic hair: Stage II (n=4) | 0
  Pubic hair: Stage III (n=4) | 0
  Pubic hair: Stage IV (n=4) | 0
  Pubic hair: Stage V (n=4) | 4
  Breast development: Stage I (n=1) | 0
  Breast development: Stage II (n=1) | 0
  Breast development: Stage III (n=1) | 0
  Breast development: Stage IV (n=1) | 0
  Breast development: Stage V (n=1) | 1

5. Secondary Outcome: Bone Age
Description: Bone age was determined by the Greulich and Pyle method using left wrist and hand X-ray.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: FAS up to Year 3: included all participants who had at least one post-baseline height measurement and were treated with the study drug for at least 1 year. Here, 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
years
  Baseline (n = 14, 15) | 8.9 [7.0 to 10.0] | 10.5 [7.0 to 13.0]
  Year 1 (n = 14, 15) | 9.5 [7.8 to 11.5] | 11.5 [7.0 to 14.0]
  Year 2 (n = 15, 13) | 10.0 [8.0 to 13.0] | 14.0 [10.0 to 14.5]
  Year 3 (n = 15, 14) | 11.3 [8.8 to 14.5] | 14.0 [11.5 to 15.0]

6. Secondary Outcome: Lean Body Mass
Description: Lean body mass, a measurement of body composition, was assessed by Dual Energy X-ray Absorptiometry (DEXA) scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: FAS up to Year 3: included all participants who had at least one post-baseline height measurement and were treated with the study drug for at least 1 year. Here, 'n' signifies those participants who were evaluable for this measure at the given time point for each group respectively.
Measure: Median (Inter-Quartile Range); unit: kilogram (kg)
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
kilogram (kg)
  Baseline (n = 15, 15) | 17.69 [14.96 to 19.96] | 23.56 [16.77 to 32.43]
  Year 1 (n = 15, 13) | 19.77 [16.62 to 24.58] | 31.16 [20.77 to 39.10]
  Year 2 (n = 14, 12) | 21.20 [18.79 to 25.13] | 34.14 [25.30 to 46.30]
  Year 3 (n = 14, 11) | 23.21 [20.88 to 25.55] | 36.38 [26.49 to 42.76]

7. Secondary Outcome: Annual Percent Change in Lean Body Mass at Year 1, 2 and 3
Description: Lean body mass, a measurement of body composition, was assessed by DEXA scan. Annual percent change: (Lean body mass at current year minus lean body mass at previous year) divided by lean body mass at previous year, multiplied by 100.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
percent change
  Annual Change at Year 1 (n = 15, 13) | 18.95 [10.04 to 21.83] | 22.97 [17.54 to 28.80]
  Annual Change at Year 2 (n = 14, 11) | 7.75 [1.31 to 12.16] | 7.33 [4.76 to 18.91]
  Annual Change at Year 3 (n = 13, 9) | 9.83 [2.67 to 13.33] | 7.90 [1.88 to 15.08]

8. Secondary Outcome: Percent Change From Baseline in Lean Body Mass at Year 3
Description: Lean body mass, a measurement of body composition, was assessed by DEXA scan. Percent change: (Lean body mass at Year 3 minus lean body mass at baseline) divided by lean body mass at baseline, multiplied by 100.
Time Frame: Baseline, Year 3
Population: FAS up to Year 3: included all participants who had at least one post-baseline height measurement and were treated with the study drug for at least 1 year. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 14 | 11
percent change | 36.82 [22.45 to 52.39] | 54.44 [43.06 to 62.30]

9. Secondary Outcome: Lean Body Mass as Percentage of Total Weight
Description: Lean body mass, a measurement of body composition, was assessed by DEXA scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percentage of total weight
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
percentage of total weight
  Baseline (n = 15, 15) | 70.56 [58.25 to 80.10] | 60.69 [55.29 to 69.14]
  Year 1 (n = 15, 13) | 76.57 [64.16 to 83.89] | 65.97 [59.58 to 76.19]
  Year 2 (n = 14, 12) | 73.32 [63.85 to 80.96] | 69.95 [59.55 to 80.07]
  Year 3 (n = 14, 11) | 72.94 [66.79 to 78.21] | 67.24 [59.83 to 74.37]

10. Secondary Outcome: Lean Body Mass Standard Deviation Score According to Chronological Age (SDS/CA)
Description: Lean body mass was assessed by DEXA scan. Lean body mass SDS/CA was obtained by measuring lean body mass, subtracting the chronological age- and gender-appropriate mean lean body mass and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 15, 15) | -1.50 [-1.81 to -0.94] | -0.90 [-1.40 to -0.54]
  Year 1 (n = 15, 13) | -1.13 [-1.64 to -0.67] | -0.52 [-0.97 to 0.20]
  Year 2 (n = 14, 12) | -1.26 [-1.94 to -0.78] | -0.87 [-1.40 to -0.32]
  Year 3 (n = 13, 11) | -1.75 [-1.96 to -0.94] | -1.29 [-2.36 to -0.14]

11. Secondary Outcome: Fat Mass
Description: Fat mass, a measurement of body composition, was assessed by DEXA scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
kg
  Baseline (n = 15, 15) | 5.47 [4.04 to 11.34] | 13.62 [9.51 to 18.05]
  Year 1 (n = 15, 13) | 4.81 [2.64 to 10.21] | 10.99 [7.22 to 18.97]
  Year 2 (n = 14, 12) | 6.97 [3.12 to 11.48] | 16.70 [5.99 to 20.59]
  Year 3 (n = 14, 11) | 6.90 [4.94 to 11.33] | 15.19 [10.28 to 22.87]

12. Secondary Outcome: Annual Percent Change in Fat Mass at Year 1, 2 and 3
Description: Fat mass, a measurement of body composition, was assessed by DEXA scan. Annual percent change: (Fat mass at current year minus fat mass at previous year) divided by fat mass at previous year, multiplied by 100.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
percent change
  Annual Change at Year 1 (n = 15, 13) | -11.21 [-24.18 to 27.46] | -3.71 [-19.44 to 15.73]
  Annual Change at Year 2 (n = 14, 11) | 29.52 [4.97 to 34.56] | -1.05 [-20.82 to 79.15]
  Annual Change at Year 3 (n = 13, 9) | 26.61 [-4.54 to 52.90] | 19.37 [10.60 to 40.12]

13. Secondary Outcome: Percent Change From Baseline in Fat Mass at Year 3
Description: Fat mass, a measurement of body composition, was assessed by DEXA scan. Percent change: (Fat mass at Year 3 minus fat mass at baseline) divided by fat mass at baseline, multiplied by 100.
Time Frame: Baseline, Year 3
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 14 | 11
percent change | 19.46 [3.83 to 73.79] | 37.56 [8.18 to 44.15]

14. Secondary Outcome: Fat Mass as Percentage of Total Weight
Description: Fat mass, a measurement of body composition, was assessed by DEXA scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percentage of total weight
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
percentage of total weight
  Baseline (n = 15, 15) | 25.0 [13.7 to 35.8] | 33.8 [29.5 to 37.2]
  Year 1 (n = 15, 13) | 17.4 [12.3 to 31.4] | 30.0 [21.9 to 34.7]
  Year 2 (n = 14, 12) | 21.1 [14.2 to 32.4] | 27.1 [15.0 to 36.2]
  Year 3 (n = 14, 11) | 21.3 [17.1 to 28.6] | 26.4 [19.1 to 37.6]

15. Secondary Outcome: Fat Mass Standard Deviation Score According to Chronological Age (SDS/CA)
Description: Fat mass was assessed by DEXA scan. Fat mass SDS/CA was obtained by measuring fat mass, subtracting chronological age- and gender-appropriate mean fat mass and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 15, 15) | 1.51 [0.50 to 2.22] | 2.20 [1.95 to 2.39]
  Year 1 (n = 15, 13) | 0.80 [-0.33 to 1.64] | 1.98 [0.88 to 2.23]
  Year 2 (n = 14, 12) | 0.86 [-0.15 to 1.66] | 1.79 [0.55 to 2.33]
  Year 3 (n = 13, 11) | 1.27 [0.25 to 1.55] | 1.74 [0.90 to 2.41]

16. Secondary Outcome: Apparent Bone Mineral Density of Lumbar Spine (BMAD [LS])
Description: BMAD (LS) was assessed by DEXA scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: gram per cubic centimeter (g/cm^3)
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
gram per cubic centimeter (g/cm^3)
  Baseline (n = 15, 14) | 0.184 [0.168 to 0.242] | 0.223 [0.211 to 0.241]
  Year 1 (n = 14, 13) | 0.209 [0.163 to 0.243] | 0.237 [0.201 to 0.244]
  Year 2 (n = 15, 14) | 0.215 [0.181 to 0.248] | 0.249 [0.217 to 0.266]
  Year 3 (n = 13, 12) | 0.239 [0.205 to 0.254] | 0.242 [0.223 to 0.266]

17. Secondary Outcome: Apparent Bone Mineral Density Standard Deviation Score of Lumbar Spine According to Chronological Age (BMAD [LS] [SDS/CA])
Description: BMAD (LS) was assessed by DEXA scan. BMAD (LS) (SDS/CA) was obtained by measuring the BMAD (LS), subtracting chronological age- and gender-appropriate mean BMAD (LS) and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 15, 14) | -3.21 [-4.02 to -1.26] | -1.53 [-1.94 to -1.35]
  Year 1 (n = 14, 13) | -2.66 [-3.70 to -1.07] | -1.51 [-2.32 to -0.95]
  Year 2 (n = 15, 14) | -2.55 [-3.74 to -0.95] | -1.42 [-1.86 to -0.72]
  Year 3 (n 12, 12) | -1.77 [-2.43 to -1.21] | -1.63 [-2.43 to -0.74]

18. Secondary Outcome: Apparent Bone Mineral Density Standard Deviation Score of Lumber Spine According to Tanner Puberty Stage (BMAD [LS] [SDS/Tanner Puberty Stage])
Description: BMAD (LS) was assessed by DEXA scan. BMAD (LS) (SDS/Tanner Puberty Stage) was obtained by measuring BMAD (LS), subtracting Tanner puberty stage- and gender-appropriate mean BMAD (LS) and dividing the result by standard deviation of that mean (as obtained from Tanner puberty stage- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 8, 8) | -4.27 [-5.47 to -2.38] | -3.09 [-3.36 to -2.31]
  Year 1 (n = 10, 7) | -3.70 [-4.80 to -2.48] | -3.23 [-4.64 to -1.74]
  Year 2 (n = 10, 9) | -4.11 [-4.36 to -1.72] | -2.60 [-3.04 to -2.17]
  Year 3 (n = 10, 8) | -3.04 [-4.06 to -2.27] | -2.96 [-3.37 to -2.76]

19. Secondary Outcome: Bone Mineral Density of Total Body (BMD [TB])
Description: BMD (TB) was assessed by DEXA scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: gram per square centimeter (g/cm^2)
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
gram per square centimeter (g/cm^2)
  Baseline (n = 15, 15) | 0.78 [0.76 to 0.86] | 0.90 [0.81 to 1.00]
  Year 1 (n = 15, 14) | 0.80 [0.76 to 0.87] | 0.92 [0.85 to 1.02]
  Year 2 (n = 14, 11) | 0.81 [0.77 to 0.89] | 0.96 [0.86 to 1.09]
  Year 3 (n = 13, 11) | 0.84 [0.80 to 0.91] | 0.99 [0.89 to 1.08]

20. Secondary Outcome: Bone Mineral Density of Lumbar Spine (BMD [LS])
Description: BMD (LS) was assessed by DEXA scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: g/cm^2
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
g/cm^2
  Baseline (n = 15, 15) | 0.55 [0.47 to 0.64] | 0.72 [0.67 to 0.85]
  Year 1 (n = 14, 14) | 0.61 [0.48 to 0.74] | 0.76 [0.66 to 0.91]
  Year 2 (n = 15, 14) | 0.64 [0.56 to 0.84] | 0.85 [0.77 to 1.04]
  Year 3 (n = 13, 12) | 0.74 [0.60 to 0.85] | 0.93 [0.79 to 1.07]

21. Secondary Outcome: Bone Mineral Content of Total Body (BMC [TB])
Description: DEXA scan of BMC was used to evaluate potential bone effects of treatment. BMC is an estimate of the amount of mineral (such as calcium) in the bone.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: gram
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
gram
  Baseline (n = 15, 15) | 636.36 [498.47 to 939.71] | 1233.58 [772.41 to 1650.08]
  Year 1 (n = 15, 14) | 775.46 [578.97 to 1119.60] | 1576.15 [939.71 to 1739.38]
  Year 2 (n = 14, 11) | 855.70 [690.07 to 1059.67] | 2003.49 [1070.42 to 2243.61]
  Year 3 (n = 13, 11) | 1112.78 [807.30 to 1176.70] | 1997.74 [1296.00 to 2195.17]

22. Secondary Outcome: Annual Percent Change in Bone Mineral Content of Total Body (BMC [TB]) at Year 1, 2 and 3
Description: BMC is an estimate of the amount of mineral (such as calcium) in the bone. Annual percent change: (BMC [TB] at current year minus BMC [TB] at previous year) divided by BMC [TB] at previous year, multiplied by 100.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
percent change
  Year 1 (n = 15, 14) | 12.51 [7.66 to 21.86] | 20.16 [11.74 to 23.05]
  Year 2 (n = 14, 11) | 17.47 [12.20 to 19.93] | 13.91 [10.63 to 18.93]
  Year 3 (n = 12, 9) | 12.03 [4.50 to 14.54] | 7.39 [7.29 to 13.30]

23. Secondary Outcome: Percent Change From Baseline in Bone Mineral Content of Total Body (BMC [TB]) at Year 3
Description: BMC is an estimate of the amount of mineral (such as calcium) in the bone. Percent change: (BMC [TB] at Year 3 minus BMC [TB] at baseline) divided by BMC [TB] at baseline, multiplied by 100.
Time Frame: Baseline, Year 3
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 13 | 11
percent change | 46.63 [24.94 to 73.91] | 60.56 [36.49 to 67.79]

24. Secondary Outcome: Bone Mineral Content Standard Deviation Score of Total Body According to Chronological Age (BMC [TB] [SDS/CA])
Description: BMC (TB) was measured by DEXA scan. BMC (TB) (SDS/CA) was obtained by measuring BMC (TB), subtracting the chronological age- and gender-appropriate mean BMC (TB) and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 15, 15) | -1.95 [-2.60 to -1.03] | -0.42 [-1.23 to 0.19]
  Year 1 (n = 15, 14) | -1.85 [-2.43 to -0.73] | -0.19 [-1.13 to 0.37]
  Year 2 (n = 14, 11) | -1.66 [-2.27 to -1.14] | -0.37 [-1.24 to 0.43]
  Year 3 (n = 12, 11) | -1.65 [-2.22 to -0.35] | -0.09 [-0.72 to 0.60]

25. Secondary Outcome: Bone Mineral Content Standard Deviation Score of Total Body According to Tanner Puberty Stage (BMC [TB] [SDS/Tanner Puberty Stage])
Description: BMC (TB) was measured by DEXA scan. BMC (TB) (SDS/Tanner Puberty Stage) was obtained by measuring BMC (TB), subtracting the Tanner puberty stage- and gender-appropriate mean BMC (TB) and dividing the result by standard deviation of that mean (as obtained from Tanner puberty stage- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 8, 8) | -2.19 [-2.47 to -0.96] | 1.41 [-0.39 to 2.46]
  Year 1 (n = 10, 8) | -1.56 [-2.24 to -0.92] | -0.52 [-1.53 to 1.65]
  Year 2 (n = 9, 7) | -2.38 [-2.72 to -1.14] | -0.47 [-1.53 to 0.37]
  Year 3 (n = 9, 7) | -2.38 [-2.56 to -1.28] | -0.17 [-1.22 to 0.83]

26. Other Pre Specified Outcome: Growth Velocity (GV)
Description: Growth velocity measures the annual rate of increase in height.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: cm/year
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
cm/year
  Baseline (n = 11, 14) | 2.9 [1.1 to 4.8] | 3.8 [2.7 to 4.4]
  Year 1 (n = 14, 15) | 6.5 [3.5 to 8.6] | 8.3 [5.4 to 8.7]
  Year 2 (n = 14, 15) | 5.3 [1.8 to 6.9] | 7.0 [4.1 to 9.2]
  Year 3 (n = 14, 14) | 4.5 [1.9 to 6.8] | 5.9 [2.3 to 7.2]

27. Other Pre Specified Outcome: Growth Velocity Standard Deviation Score According to Chronological Age (GV [SDS/CA])
Description: GV measures the annual rate of increase in height. GV (SDS/CA) was obtained by measuring GV, subtracting the chronological age- and gender-appropriate mean GV and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 10, 14) | -1.7 [-2.8 to -1.3] | -2.2 [-2.9 to -1.3]
  Year 1 (n = 14, 15) | 1.0 [-1.5 to 3.9] | 1.3 [-0.7 to 1.9]
  Year 2 (n = 14, 15) | 0.1 [-1.9 to 3.7] | 2.9 [1.4 to 4.2]
  Year 3 (n = 14, 14) | 0.4 [-0.5 to 2.1] | 2.9 [-0.1 to 5.7]

28. Other Pre Specified Outcome: Growth Velocity Standard Deviation Score According to Bone Age (GV [SDS/BA])
Description: GV measures the annual rate of increase in height. GV (SDS/BA) was obtained by measuring GV, subtracting the bone age- and gender-appropriate mean GV and dividing the result by standard deviation of that mean (as obtained from bone age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: SDS
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
SDS
  Baseline (n = 9, 14) | -2.8 [-3.9 to -1.7] | -2.1 [-2.4 to -1.1]
  Year 1 (n = 13, 15) | 0.8 [-0.9 to 2.9] | 0.6 [-0.6 to 2.4]
  Year 2 (n = 14, 13) | -0.3 [-3.9 to 1.1] | 1.4 [-0.6 to 2.0]
  Year 3 (n = 14, 14) | -0.9 [-2.2 to 0.9] | 0.1 [-1.7 to 3.4]

29. Other Pre Specified Outcome: Insulin-like Growth Factor-1 (IGF-1) Concentration up to Year 3
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome)
Number analyzed (Participants) | 15 | 15
nanogram per milliliter (ng/mL)
  Baseline (n = 15, 12) | 157.0 [61.0 to 345.0] | 344.5 [191.0 to 719.0]
  Year 1 (n = 15, 15) | 400.0 [154.0 to 1370] | 952.0 [424.0 to 1658.0]
  Year 2 (n = 15, 14) | 388.0 [188.0 to 1338.0] | 880.0 [311.0 to 1718.0]
  Year 3 (n = 15, 14) | 405.0 [239.0 to 1160.0] | 657.0 [323.0 to 1298.0]

30. Other Pre Specified Outcome: Insulin-like Growth Factor-1 (IGF-1) Concentration After Year 3
Time Frame: Year 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10; 0.5 and 1 year after somatropin discontinuation, Final Height (assessed up to Year 11)
Population: FAS After year 3: included all participants who received at least 1 dose of the study treatment and who had at least 1 post-baseline height measurement. Here, 'n' signifies those participants who were evaluable for this measure at given time point.
Measure: Median (Full Range); unit: milligram per deciliter (mg/dL)
Arm/Group | Somatropin- After Year 3
Number analyzed (Participants) | 21
milligram per deciliter (mg/dL)
  Year 3.5 (n = 8) | 0.05 [0.04 to 0.09]
  Year 4 (n = 19) | 0.06 [0.03 to 0.10]
  Year 4.5 (n = 16) | 0.06 [0.02 to 0.14]
  Year 5 (n = 17) | 0.05 [0.02 to 0.09]
  Year 5.5 (n = 11) | 0.06 [0.02 to 0.09]
  Year 6 (n = 14) | 0.05 [0.02 to 0.08]
  Year 6.5 (n = 8) | 0.07 [0.02 to 0.09]
  Year 7 (n = 8) | 0.06 [0.02 to 0.07]
  Year 7.5 (n = 4) | 0.05 [0.03 to 0.07]
  Year 8 (n = 6) | 0.06 [0.03 to 0.07]
  Year 8.5 (n = 2) | 0.08 [0.07 to 0.08]
  Year 9 (n = 2) | 0.06 [0.06 to 0.07]
  Year 9.5 (n = 1) | 0.07 [0.07 to 0.07]
  Year 10 (n = 1) | 0.05 [0.05 to 0.05]
  0.5 years after somatropin discontinuation (n = 2) | 0.03 [0.03 to 0.04]
  1 year after somatropin discontinuation (n = 2) | 0.03 [0.02 to 0.05]
  Final height (n = 3) | 0.06 [0.05 to 0.07]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) | Somatropin- Up To Year 3 (Nephrotic Syndrome) | Somatropin- After Year 3
Serious Adverse Events (participants affected / at risk) | 13/15 | 14/15 | 19/21
Other Adverse Events (participants affected / at risk) | 13/15 | 14/15 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) (N=15) | Somatropin- Up To Year 3 (Nephrotic Syndrome) (N=15) | Somatropin- After Year 3 (N=21)
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Biopsy kidney (Investigations) | 0 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0
Condition aggravated (General disorders) | 3 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 2
Disease recurrence (General disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Insulin resistant diabetes (Metabolism and nutrition disorders) | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 6
Nephrotic syndrome (Renal and urinary disorders) | 0 | 9 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Keratopathy (Eye disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 3
Headache and abdominal pain (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin- Up To Year 3 (Juvenile Idiopathic Arthritis) (N=15) | Somatropin- Up To Year 3 (Nephrotic Syndrome) (N=15) | Somatropin- After Year 3 (N=21)
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 2
Auricular perichondritis (Ear and labyrinth disorders) | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2
Face oedema (General disorders) | 1 | 0 | 1
Hyperthermia (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 2 | 2
Bronchitis (Infections and infestations) | 1 | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 3 | 2
Gastroenteritis (Infections and infestations) | 0 | 2 | 3
Influenza (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 3 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 3 | 2
Tracheobronchitis (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 2
Viral tracheitis (Infections and infestations) | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Insulin-like growth factor increased (Investigations) | 0 | 3 | 3
Red blood cell sedimentation rate increased (Investigations) | 5 | 0 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Sodium retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Joint effusion (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 5
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 3
Depression (Psychiatric disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Hypercalciuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 11 | 7
Proteinuria (Renal and urinary disorders) | 0 | 6 | 3
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood human immunodeficiency virus (HIV) ribo-nucleic acid (RNA) increased (Investigations) | 0 | 0 | 1
Blood follicle stimulating hormone increased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 3
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 4
Mineral deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bronchopneumopathy due to mycoplasm's infection (General disorders) | 0 | 0 | 1
Fever, rhynopharyngal infection, macular exenthema and Asthenia (General disorders) | 0 | 0 | 1
Ocular hypertony (General disorders) | 0 | 0 | 1
Uremic rectal bleeding (pratouayia) (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Results for secondary and other pre-specified endpoints (except IGF-1) are reported for only up to 3 years because data beyond Year 3 was not summarized as the study was terminated due to Good Clinical Practice (GCP) non-compliance issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.